CLINICAL TRIAL: NCT02088619
Title: Positive Psychotherapy to Improve Autonomic Function and Mood in ICD Patients
Brief Title: Positive Therapy for Autonomic Function & Mood in ICD Patients
Acronym: PAM-ICD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00028869; 1R34HL107733-01A1 (NIH)
Record Dates: First submitted 2014-02-18; First posted 2014-03-17 (Estimated); Last update posted 2017-10-02 (Actual); Status verified 2017-09

CONDITIONS: Ventricular Arrhythmia; Implantable Cardioverter Defibrillator
Keywords: psychological wellbeing; anxiety; depression; autonomic functioning
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Quality of Life Therapy (QOLT) (Experimental): Positive emotion-focused cognitive behavioral psychotherapy
  Interventions: Behavioral: Quality of Life Therapy (QOLT)
- Heart Healthy Education (HHE) (Active Comparator): Heart healthy education program
  Interventions: Behavioral: Heart Healthy Education (HHE)

INTERVENTIONS:
Behavioral: Quality of Life Therapy (QOLT)
  Arms: Quality of Life Therapy (QOLT)
Behavioral: Heart Healthy Education (HHE)
  Arms: Heart Healthy Education (HHE)

SUMMARY:
The purpose of this 2-group randomized clinical trial is to: 1) examine the feasibility and acceptability of a 3-month positive-emotion focused therapy (Quality of Life Therapy) modified specifically for patients with implantable cardioverter defibrillator (ICD); and 2) obtain estimates of effect size for QOLT compared to Heart Healthy Education on the changes in arrhythmia frequency and biomarkers of autonomic function, as well as changes in emotion, mood, and well-being across time (baseline, 3 & 9-months). It is hypothesized that the QOLT will promote improvements in autonomic function, reduced arrhythmia frequency, and improved psychological well-being.

ELIGIBILITY:
Inclusion Criteria:

1. Adult men and women (≥18 years of age) who have received an ICD for primary or secondary prevention of sudden cardiac death. All patients will have systolic left ventricular dysfunction due to coronary disease or nonischemic cardiomyopathy. There is no requirement for time since implant;
2. Score ≥5 on the Hospital Anxiety and Depression Scale (HADS) anxiety or depression scales;
3. Able to read and write English
4. Able to commit to the 3-month QOLT/HHE program and 3 assessments over a 9-month duration.

Exclusion Criteria:

1. >5% atrial or ventricular pacing;
2. Sinus node dysfunction;
3. Persistent and permanent atrial fibrillation (AF) (h/o of paroxysmal AF will be allowed).
4. Long QT syndrome; and other channelopathies such as Brugada syndrome;
5. Hypertrophic cardiomyopathy;
6. Neurocognitive or cognitive impairments;
7. Severe psychopathology that warrants intensive treatment;
8. Participation in another research trial; and
9. Currently in psychological or psychiatric treatment.
10. Current psychotropic and cardiac medication prescriptions and usage need to be stable (i.e., no change in type or dosage) for 3-months prior to study enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Frequency of arrhythmias between baseline and 3-months | 3-months
  Total arrhythmia frequencies between baseline and 3-months will be the sum of non-sustained ventricular tachycardia (NSVT) detected on the Holter ( ≥6 beats, at >120 beats per minute [BPM] ) plus arrhythmias detected by the ICD
Frequency of arrhythmias between 3-months and 9-months | 9-months
  Total arrhythmia frequencies between 3-months and 9-months will be the sum of non-sustained ventricular tachycardia (NSVT) detected on the Holter ( ≥6 beats, at >120 BPM ) plus arrhythmias detected by the ICD

SECONDARY OUTCOMES:
Frequency of ICD therapies between baseline and 3-months | 3-months
  Obtained from ICD interrogation reports from recording between baseline and 3-months
Change in High Frequency heart rate variability (HF-HRV) between baseline and 3-months | 3-months
  Index of parasympathetic activity; obtained from 24-hour Holter recording
Frequency of ICD therapies between 3-months and 9-months | 9-months
  Obtained from ICD interrogation reports between 3- and 9-months
Change in High Frequency heart rate variability (HF-HRV) between 3- and 9-months | 9-months
  Index of parasympathetic activity; obtained from 24-hour Holter recording

OTHER OUTCOMES:
Florida Shock Anxiety Scale | 3 months
Florida Patient Acceptance Scale | 3-months
Emotions Questionnaire | 3-months
Center for Epidemiologic Studies - Depression Scale (CES-D) | 3-months
State Trait Anxiety Inventory (STAI) | 3-months
Life Orientation Test - Revised (LOT-R) | 3-months
Positive and Negative Affect Schedule (PANAS) | 3-months
Satisfaction with Life Scale (SWLS) | 3-months
Quality of Life Inventory (QOLI) | 3-months
Short-Form Health Survey-36 (SF-36) | 3-months
Minnesota Living with Heart Failure Questionnaire (MLHFQ) | 3-months

CONTACTS AND LOCATIONS:
Overall Officials: Eva R Serber, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Dept of Psychiatry, Division of Bio-Behavioral Medicine, Charleston, South Carolina, United States

REFERENCES:
- [Background] Frisch M. Quality of Life Therapy; Applying a Life Satisfaction Approach to Positive Psychology and Cognitive Therapy. Hobokon, NJ: John Wiley & Sons, Inc.; 2006.